CLINICAL TRIAL: NCT04274465
Title: Application of Plasma Circulating Human Papillomavirus (HPV) DNA Testing to Management of Cervical Intraepithelial Neoplasia
Brief Title: Application of Plasma Circulating HPV DNA Testing to Management of Cervical Intraepithelial Neoplasia
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1928
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cervix Lesion; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue collected will be retained for 15 years and will be tested for cHPVDNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Negative high risk (HR)-HPV, cytology co-test
  Interventions: Diagnostic Test: digital PCR (dPCR) assay
- CIN 1: Biopsy with low grade dysplasia
  Interventions: Diagnostic Test: digital PCR (dPCR) assay
- CIN 2-3: Biopsy with high grade dysplasia
  Interventions: Diagnostic Test: digital PCR (dPCR) assay

INTERVENTIONS:
Diagnostic Test: digital PCR (dPCR) assay — It is a highly sensitive and specific droplet digital PCR assay for absolute quantification of circulating tumor HPV DNA for the most prevalent HPV types that will determine if a woman has cHPVDNA

SUMMARY:
The purpose of this study is to see if circulating HPV DNA (cHPVDNA) can be used as a noninvasive biomarker for cervical intraepithelial neoplasia (CIN) 2-3 in hopes of reducing procedures and costs for patients, as well as personalize their treatment plan.

DETAILED DESCRIPTION:
cHPVDNA is detectable in plasma of patients with invasive disease and CIN 1-3, and with the development of a highly sensitive and specific droplet digital Polymerase Chain Reaction (PCR) assay, it is hoped to be identified more prevalently and thus can improve risk stratification and help produce personalized treatment decisions and may be more cost-efficient. Plasma samples and cervical swabs will be collected from patients in University of North Carolina (UNC) Gynecology clinics, and some patients will also provide a urine sample. Those receiving biopsies or colposcopies and will come back to clinic 2-4 weeks post-excision for collection of another blood specimen. Using plasma samples and pathology results, we will characterize the relationship between plasma cHPVDNA levels and 1) CIN 1 versus CIN 2-3 pathology 2) CIN 2-3 pre-excision and 2-4 weeks post-excision. We will accrue three cohorts of 25, 30, 30 patients corresponding to 1) Control 2) CIN 1 3) CIN 2-3. The control cohort will establish background signal in the assay. We will compare the proportion of detectable cHPVDNA levels between CIN 1 and CIN 2-3 cohorts using Fisher's exact test with 80% power, significance level of 10%. Paired t-test will be used to compare pre- and post-excision cHPVDNA levels.

ELIGIBILITY:
Inclusion Criteria:

* No history of previously treated cervical cancer
* Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee

Exclusion Criteria:

* Women who are pregnant or nursing

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women ≥ 18 years old who are presenting to UNC Gynecology clinics with or without dysplasia and may or may not need colposcopy, biopsy, or lesion excisions.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Relationship between plasma cHPVDNA levels and presence of CIN 2-3 histopathology | Baseline
  We will quantify cHPVDNA levels in blood plasma from patients with normal screening, CIN 1, and CIN 2-3 cervical disease prior to treatment.

SECONDARY OUTCOMES:
Changes in cHPVDNA levels following excisional therapy for CIN 2-3 cervical disease. | 2-4 weeks post-excision
  For patients who undergo excisional therapy, we will collect bio-specimens and quantify cHPVDNA levels in plasma during their post-procedure visit.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sud, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Tuvara Jenene King, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials